CLINICAL TRIAL: NCT05314335
Title: The Effect of Reflexology Socks On The Management of Opioid-Induced Constipation
Brief Title: Reflexology Socks and Opioid-induced Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Ferda AKYUZ OZDEMIR, MsCN, Research Assistant, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FAKYUZOZDEMİR
Record Dates: First submitted 2022-03-18; First posted 2022-04-06 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Opioid Use; Constipation; Reflexology
Keywords: Opioid induced Constipation; Reflexology
MeSH Terms: conditions — Constipation; Opioid-Induced Constipation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reflexology socks+Walking (Experimental): In the first interview; patient diagnosis form and Constipation Quality of Life scale will be applied. In order to evaluate the routine bowel habits of the patients, no application will be made in the first week and the patients will be asked to complete the Defecation Diary, Visual Comparison Scale and the Bristol Stool Consistency Scale for 1 week when defecation occurs. Afterwards, the reflexology socks designed by the researcher for the patients; will be told to wear and walk 30 minutes after breakfast and dinner for 30 minutes 3 days a week (Monday, Wednesday and Friday). Patients will be asked to continue the application for 4 weeks. The patients will be administered the Defecation Diary, the Visual Comparison Scale, and the Bristol Stool Consistency Scale when defecation occurs daily during the application. In addition, on the 30th day of the application, the Constipation Quality of Life Scale will be administered to the patients again.
  Interventions: Other: Reflexology socks+walking
- Just walking (Other): In the first interview, patient diagnosis form and Constipation Quality of Life scale will be applied. In order to evaluate the routine bowel habits of the patients, no application will be made in the first week and the patients will be asked to complete the Defecation Diary, Visual Comparison Scale and the Bristol Stool Consistency Scale for 1 week when defecation occurs. Subsequently, patients will be instructed to walk for 30 minutes, 3 days a week (Monday, Wednesday, and Friday), 30 minutes after breakfast and dinner. Patients will be asked to continue the application for 4 weeks. The patients will be administered the Defecation Diary, the Visual Comparison Scale and the Bristol Stool Consistency Scale when defecation occurs daily during the application. In addition, on the 130th day of the application, the Constipation Quality of Life Scale will be administered to the patients again.
  Interventions: Other: Just walking

INTERVENTIONS:
Other: Reflexology socks+walking — Patients should wear reflexology socks; Wearing clothes and walking 30 minutes after breakfast and dinner for 30 minutes 3 days a week (Monday, Wednesday and Friday)
  Arms: Reflexology socks+Walking
Other: Just walking — Patients will be instructed to walk for 30 minutes, 3 days a week (Monday, Wednesday, and Friday), 30 minutes after breakfast and dinner. Patients will be asked to continue the application for 4 weeks.
  Arms: Just walking

SUMMARY:
Opioids are one of the most commonly used treatment approaches in the treatment of severe pain due to cancer and non-cancer causes. The most commonly reported side effect by patients related to opioid use is constipation. Opioid-related constipation, with an overall incidence of between 17% and 88%, requires a reduction in the treatment dose or drug rotation in some patients. It also makes it difficult for patients to comply with treatment. However, if the constipation due to opioid use is not managed properly and continues for a long time, many problems such as hemorrhoids and perforation, rectal pain and burning, intestinal rupture, anal fissure, diarrhea due to partial obstruction, urinary incontinence may develop.

It is known that reflexology application applied to the foot increases parasympathetic activity while inhibiting sympathetic activity. Peristalsis and bowel movements are reduced in patients with opioid-related constipation. Reflexology practice; It is thought that an increase in motility can be achieved by increasing parasympathetic activity. However, it is thought that the development of reflexology socks will be more effective due to the difficulties of finding a reflexology specialist, the difficulty of reaching a reflexology specialist and the difficulty of having them applied at home. Thanks to the insoled reflexology socks, which have silicone balls that apply pressure to the stomach, liver, small intestine, large intestine and solar plexus points, patients will be able to wear them easily at home and perform their daily life activities at the same time. It is thought that reflexology stockings can be effective in reducing opioid-related constipation, together with being inexpensive and easy to apply.

The aim of this study is to examine whether reflexology stockings are an effective approach in reducing opioid-related constipation.

DETAILED DESCRIPTION:
The basis of the physiopathological mechanism of constipation due to opioid use is the reducing effect on intestinal motility. There are opioid receptors called "mu" in the enteric nervous system. In patients using opioids, opioid agonists bind to these receptors. As a result of the binding of opioid agonists to the "mu" receptors, the release of excitatory and inhibitory neurotransmitters is inhibited and the coordinated rhythmic contractions required for bowel movements are reduced, as a result, peristaltic movements in the ileum and colon slow down and opioid-related intestinal dysfunction develops. With the prolonged stay of feces in the intestinal lumen, fluid absorption from the intestine increases and dry, hard stools are formed. Sphincter tone and non-impulsive contractions increase. As a result of all these effects, constipation develops.

In the management of constipation; In this study, both the effects of reflexology applied to the foot on the neuropeptide system and the effect of regulating electromagnetic transmissions were utilized. In a study conducted with the participation of children with cerebral palsy with constipation, it was reported that reflexology applied to the foot twice a week for 8 weeks had a positive effect on constipation. In a different study evaluating the effect of foot reflexology in patients with Multiple Sclerosis, it was reported that reflexology massage applied to the stomach, liver, small intestine, large intestine and solar plexus points for 30-40 minutes once a week for 6 weeks reduced constipation. In a different study conducted with the participation of elderly patients, it was reported that foot reflexology applied to the stomach, liver, small intestine, large intestine and solar plexus points for 30 minutes 3 times a week for 1 month resulted in a significant increase in bowel movements. In a systematic review and meta-analysis study evaluating the effect of foot reflexology in the management of functional constipation; It has been concluded that foot reflexology has a positive effect on stool frequency, stool consistency, difficult defecation, incomplete emptying of the intestines, abdominal pain and bloating. However, since the randomized controlled studies included in this study were studies with small sample groups, it was stated that larger studies were needed.

In addition to the effects in these studies, it is known that reflexology application applied to the foot increases parasympathetic activity while inhibiting sympathetic activity. Peristalsis and bowel movements are reduced in patients with opioid-related constipation. Reflexology practice; It is thought that an increase in motility can be achieved by increasing parasympathetic activity. However, it is thought that the development of reflexology socks will be more effective due to the difficulties of finding a reflexology specialist, the difficulty of reaching a reflexology specialist and the difficulty of having them applied at home. Thanks to the insoled reflexology socks, which have silicone balls that apply pressure to the stomach, liver, small intestine, large intestine and solar plexus points, patients will be able to wear them easily at home and perform their daily life activities at the same time. It is thought that reflexology stockings can be effective in reducing opioid-related constipation, together with being inexpensive and easy to apply.

RESEARCH PROTOCOL The patients will be divided into 2 groups as experimental and control groups according to the predetermined randomization control list. In the first interview with the patients in the experimental group; patient diagnosis form and Constipation Quality of Life scale will be applied. In order to evaluate the routine bowel habits of the patients, no application will be made in the first week and the patients will be asked to complete the Defecation Diary, Visual Comparison Scale and the Bristol Stool Consistency Scale for 1 week when defecation occurs. Afterwards, the reflexology socks designed by the researcher for the patients; will be told to wear and walk 30 minutes after breakfast and dinner for 30 minutes 3 days a week (Monday, Wednesday and Friday). Patients will be asked to continue the application for 4 weeks. The patients will be administered the Defecation Diary, the Visual Comparison Scale, and the Bristol Stool Consistency Scale when defecation occurs daily during the application. In addition, on the 15th and 30th days of the application, the Constipation Quality of Life Scale will be administered to the patients again.

For the patients in the control group; In the first interview, patient diagnosis form and Constipation Quality of Life scale will be applied. In order to evaluate the routine bowel habits of the patients, no application will be made in the first week and the patients will be asked to complete the Defecation Diary, Visual Comparison Scale and the Bristol Stool Consistency Scale for 1 week when defecation occurs. Subsequently, patients will be instructed to walk for 30 minutes, 3 days a week (Monday, Wednesday, and Friday), 30 minutes after breakfast and dinner. Patients will be asked to continue the application for 4 weeks. The patients will be administered the Defecation Diary, the Visual Comparison Scale, and the Bristol Stool Consistency Scale when defecation occurs daily during the application. In addition, on the 15th and 30th days of the application, the Constipation Quality of Life Scale will be administered to the patients again.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are at least 18 years old ( ≥ 18 years old)
* Patients with a maximum age of 85 years (≤ 85 years old)
* Patients who volunteered to participate in the study
* Does not have any disability in communicating cognitively, mentally and verbally.
* Opioid treatment applied for approximately 2 weeks
* Those with constipation complaints
* At least one of the constipation problems (straining during bowel emptying, hard stool, feeling of incomplete evacuation, gas/bloating, rectal pressure/defecation sensation) that have been emptied less than 3 times a week since the opioid treatment started and/or developed due to opioid use patients
* Patients with a foot number between 37-44

Exclusion Criteria:

* Having a complaint of peripheral neuropathy
* Being diagnosed with diabetes
* Having impaired skin integrity
* Having any deformity of flat feet or feet

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
The change in defecation routine ( frequency, amount of stool etc.) | Every day / for 5 weeks
  The daily defecation routine of the patients was assessed with the Daily Defecation Scale. With this chart, the amount of stool, stool consistency, straining during defecation, feeling of incomplete evacuation after defecation, and number of defecations are monitored weekly. With this form, patients recorded their defecation status for 5 weeks each time they defecated. Scores collected for each symptom of constipation are calculated by dividing the number of defecations in the same week.
The change in the severity of the symptoms of constipation | Every day / for 5 weeks
  The changes in constipation-related symptoms were assessed with the Visual Comparison Scale.
  Visual Comparison Scale: It is a 6-question scale that evaluates the severity of the symptoms of constipation (constipation severity, straining, feeling of incomplete evacuation, rectal fullness, rectal pain and gas) in the patient. The visual comparison scale consists of a horizontal line between 0-10.
The change in stool consistency and type. | At the time of defecation/ for 5 weeks
  At the time of defecation, stool consistency and type were assessed with the Bristol Stool Scale.This scale is used to evaluate stool shape and form in order to monitor changes in bowel functions. Stool shape is classified into 7 different categories. In this scale, which accepts that the stool form changes with the residence time of the stool in the colon; 1 and 2 type patients have Constipation, 3 and 4 types have normal stools and 5-7. type indicates that the patient has diarrhea.
The change in quality of life due to constipation | At baseline, at day 15 and at day 30.
  The change in quality of life due to constipation was assessed with the Constipation Quality of Life Scale.
  Constipation Quality of Life Scale: The item scores of this Likert-type scale range from 1 to 5. The subscales of this 28-item scale are "Anxiety/Anxiety" (11 items), "Physical Discomfort" (4 items), "Psychosocial Discomfort" (8 items), "Satisfaction" (5 items).

CONTACTS AND LOCATIONS:
Overall Officials: Ferda AKYÜZ ÖZDEMİR, Principal Investigator — Mugla Sıtkı Koçman University Fethiye Faculty of Health Sciences
Locations (1):
- Mugla Sitki Kocman University, Fethiye, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No